CLINICAL TRIAL: NCT05211622
Title: OZOCLO: a Randomized Clinical Trial for Prevention of Oral Mucositis
Brief Title: OZOCLO_MUCOSITIS: a New Protocol for Prevention of Oral Mucositis
Acronym: OZOCLO_MUCOS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Olga Di Fede, Associate Professor, University of Palermo
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: OZOCLO_MUCOSITIS 01_2021
Record Dates: First submitted 2021-12-14; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2021-12

CONDITIONS: Mucositis (MeSH Unique ID: D052016); Stomatitis (MeSH Unique ID: D013280)
MeSH Terms: conditions — Mucositis; Stomatitis | interventions — Sodium Bicarbonate

STUDY DESIGN:
Intervention Model Description: Patients will be randomly using a table of random numbers (allocation ratio 1:1:1:1).
  * Arm I, OZOCLO
    1. alpha acid lipoic - 600 mg/die per os from 7 days before the beginning of chemotherapy and for other 4 die
    2. ozonated oil - mouthwash (1 minute- three times/die) for 2 weeks
    3. chlorhexidine 0,2% - mouthwash (1 minute- three times/die) from five days after the beginning and for other 2 weeks
  * Arm II, OBC Sodium bicarbonate 5% solution - mouthwash (1 minute- three times/die) for 3 weeks
  * Arm III, CHX Chlorhexidine 0,2% - mouthwash (1 minute- three times/die) from five days after the beginning and for other 2 weeks
  * Arm IV, AAL-OZ
    1. alpha acid lipoic - 600 mg/die per os from 7 days before the beginning and continue for other 4 die
    2. ozonated oil - mouthwash (1 minute- three times/die) from the beginning and for 2 weeks Every interventional arm will be conducted by the patient at home according to indications and will monitored at 8th, 15th, and the 21st day
Who Masked: Participant, Investigator
Masking Description: Nobody else
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group I, OZOCLO (Experimental): • Group I, OZOCLO
  1. alpha acid lipoic - 600 mg/die per os from 7 days before the beginning of chemotherapy and continue for other 4 days
  2. ozonated oil - mouthwash (1 minute- three times/die after oral hygiene, possibly) from the beginning of chemotherapy and for 2 weeks
  3. chlorhexidine 0,2% - mouthwash (1 minute- three times/die after oral hygiene, possibly) from five days after the beginning of chemotherapy and for subsequent 2 weeks
  Interventions: Drug: 1. alpha acid lipoic - tables; Drug: 2. ozonated oil - mouthwash; Drug: 3. chlorhexidine 0,2% - mouthwash
- Group II, OBC (Placebo Comparator): • Group II, OBC Sodium bicarbonate 5% solution - mouthwash (1 minute- three times/die after oral hygiene, possibly) from the beginning of chemotherapy and for 3 weeks
  Interventions: Drug: 4. sodium bicarbonate 5% solution - mouthwash
- Group III, CHX (Active Comparator): • Group III, CHX Chlorhexidine 0,2% - mouthwash (1 minute- three times/die after oral hygiene, possibly) from five days after the beginning of chemotherapy and for subsequent 2 weeks
  Interventions: Drug: 3. chlorhexidine 0,2% - mouthwash
- Group IV, AAL-OZ (Active Comparator): • Group IV, AAL-OZ
  1. alpha acid lipoic - 600 mg/die per os from 7 days before the beginning of chemotherapy and continue for other 4 days
  2. ozonated oil - mouthwash (1 minute- three times/die after oral hygiene, possibly) from the beginning of chemotherapy and for 2 weeks
  Interventions: Drug: 1. alpha acid lipoic - tables; Drug: 2. ozonated oil - mouthwash

INTERVENTIONS:
Drug: 1. alpha acid lipoic - tables — 600 mg/die per os from 7 days before the beginning of chemotherapy and continue for other 4 days
  Other Names: alpha acid lipoic - tables
  Arms: Group I, OZOCLO; Group IV, AAL-OZ
Drug: 2. ozonated oil - mouthwash — 1 minute- three times/die after oral hygiene, possibly, from the beginning of chemotherapy and for 2 weeks
  Other Names: ozonated oil - mouthwash
  Arms: Group I, OZOCLO; Group IV, AAL-OZ
Drug: 3. chlorhexidine 0,2% - mouthwash — 1 minute- three times/die after oral hygiene, possibly, from five days after the beginning of chemotherapy and for subsequent 2 weeks
  Other Names: chlorhexidine 0,2% - mouthwash
  Arms: Group I, OZOCLO; Group III, CHX
Drug: 4. sodium bicarbonate 5% solution - mouthwash — 1 minute- three times/die after oral hygiene, possibly, from the beginning of chemotherapy and for 3 weeks
  Other Names: sodium bicarbonate 5% solution - mouthwash
  Arms: Group II, OBC

SUMMARY:
Oral mucositis (OM) is a significant side effect of cytotoxic anti-cancer chemotherapy and HN radiotherapy. CT-associated OM (CT-OM). It is the ulcerative phase that is most painful and associated with poor health outcomes. The sequelae of CT-OM, which include pain, odyno/dys-phagia, dysgeusia, decreased oral intake and systemic infection, frequently require treatment delays, interruptions, and discontinuations that not only negatively impact the quality of life but also tumor control and survivorship. To date, OM management is aimed to control symptoms through topical or systemic analgesics and topical application of barrier agents to cover injured mucosa as a salve or ointment. According to the recent MASCC/ISOO Clinical Practice Guidelines for the Management of Mucositis Secondary to Cancer Therapy, no guideline was possible regarding the use of saline or sodium bicarbonate rinses in the prevention or treatment of OM-CT in patients undergoing cancer therapy because of limited data.

Ozone at low medical concentration, not included in MASCC guidelines, will be generally proven to induce a mild activation of protective anti-oxidant pathways, thus exerting therapeutic effects in many inflammatory diseases.

Aim: to evaluate the effectiveness of a new protocol OZOCLO (alpha-lipoic acid, ozonated oil, and chlorhexidine [CHX] mouthwash) compared to sodium bicarbonate solution (Oral Basic Care- OBC) or chlorhexidine (CHX) mouthwash alone or to a binomial administration (AAL-OZ) of systemic alpha-lipoic acid and topical ozonated oil to reduce the incidence of OM (primary aim) and/or to postpone the beginning of oral mucositis (OM) and to reduce OM severity (secondary aims).

DETAILED DESCRIPTION:
Oral mucositis (OM) is a significant side effect of cytotoxic anti-cancer chemotherapy and HN radiotherapy. CT-associated OM (CT-OM) begins in the submucosa and becomes clinically on the surface about 4 days after infusion: typical primary manifestations are erythema, mucosal atrophy, and sensitivity. The process continues to deteriorate mucosae, and ulceration occurs a few days later, peaking at 2 weeks and persisting for 1-2 weeks after which it typically resolves spontaneously. It is the ulcerative phase that is most painful and associated with poor health outcomes. The sequelae of CT-OM, which include pain, odyno/dys-phagia, dysgeusia, decreased oral intake and systemic infection, frequently require treatment delays, interruptions, and discontinuations that not only negatively impact the quality of life but also tumor control and survivorship. To date, OM management is aimed to control symptoms through topical or systemic analgesics and topical application of barrier agents to cover injured mucosa as a salve or ointment. Although the investigators reviewed a large body of evidence, there are still, clinical settings for which there is no recommended intervention. According to the recent MASCC/ISOO Clinical Practice Guidelines for the Management of Mucositis Secondary to Cancer Therapy, no guideline was possible regarding the use of saline or sodium bicarbonate rinses in the prevention or treatment of OM-CT in patients undergoing cancer therapy because of limited data. Despite the limited data available for both saline and sodium bicarbonate, the panel recognizes that these are inert, bland rinses that increase oral clearance, which may help maintain oral hygiene and improve patient comfort. Also, CHX is indicated because of concurrent oral infection and OM, it is acceptable to use it for the oral infection.

Ozone at low medical concentration, not included in MASCC guidelines, will be generally proven to induce a mild activation of protective anti-oxidant pathways, thus exerting therapeutic effects in many inflammatory diseases.

Aim: to evaluate the effectiveness of a new protocol OZOCLO (alpha-lipoic acid, ozonated oil, and chlorhexidine [CHX] mouthwash) compared to sodium bicarbonate solution (Oral Basic Care- OBC) or chlorhexidine (CHX) mouthwash alone or to a binomial administration (AAL-OZ) of systemic alpha-lipoic acid and topical ozonated oil to reduce the incidence of OM (primary aim) and/or to postpone the beginning of oral mucositis (OM) and to reduce OM severity (secondary aims).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80 years
* Planned to receive conventional chemotherapy such as:

  * CMF (cyclophosphamide (Endoxan), methotrexate, 5-FU))
  * Standard AC+T regimen (doxorubicin (Adriamycin)), cyclophosphamide (Endoxan), Taxane [paclitaxel (Taxol) or docetaxel (Taxotere)) or any combination of two or more components (e.g., ACT, TAC, TA, AT, AC)
  * ABVD (doxorubicin (Adriamycin), bleomycin, vinblastine, dacarbazine)
  * FOLFIRI (irinotecan, 5-FU, leucovorin)
  * Any other 5-FU-based regimen
* Planned to receive at conventional new generation targeted agents (tyrosine-kinase inhibitors or monoclonal antibodies) such as cetuximab, axitinib, bevacizumab, sunitinib, and sorafenib, temsirolimus, everolimus, vemurafenib, dabrafenib.
* Be willing and able to complete all study-related activities
* Properly obtained written informed consent

Exclusion Criteria:

* Receiving any oxaliplatin-containing chemotherapy regimen, such as FOLFOX
* Concurrent radiotherapy
* Unable or unwilling to complete study assessments
* Concurrent participation in another interventional clinical study or use of another investigational agent within 30 days before randomization
* Any other clinical or psychiatric condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the protocol
* Chronic use of opioid analgesics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-03-10 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-10 (Estimated)

PRIMARY OUTCOMES:
Change of OM incidence | 7th, 14th, and the 21st day after application of the interventions
  In order to demonstrate whether the new protocol OZOCLO determines change of the incidence of OM compared to sodium bicarbonate solution (OBC) or chlorhexidine (CHX) mouthwash alone or the binomial AAL-OZ combination, in patients treated with chemotherapy regimens.

SECONDARY OUTCOMES:
Delay onset of OM | 7th, 14th, and the 21st day after application of the interventions
  In order to determine whether the new protocol OZOCLO determines a delay of onset for OM, considering that it currently begins at 7th day, compared to sodium bicarbonate solution (OBC) or chlorhexidine (CHX) mouthwash alone or a binomial administration of systemic alpha-lipoic acid and topical ozonated oil.

OTHER OUTCOMES:
OM severity assessment | 7th, 14th, and the 21st day after application of the interventions
  To reduce OM severity, assuming one-point score difference (assessed through the Oral Mucositis World Health Organization Toxicity Scale- from grade 0 - none to grade IV- Oral alimentation impossible) compared to chlorhexidine (CHX) mouthwash alone or a binomial administration of systemic alpha-lipoic acid and topical ozonated oil and two-point score difference compared to sodium bicarbonate solution at one year.

CONTACTS AND LOCATIONS:
Overall Officials: Olga Di Fede, Professor, Principal Investigator — University of Palermo, Di.Chir.On.S

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Elad S, Cheng KKF, Lalla RV, Yarom N, Hong C, Logan RM, Bowen J, Gibson R, Saunders DP, Zadik Y, Ariyawardana A, Correa ME, Ranna V, Bossi P; Mucositis Guidelines Leadership Group of the Multinational Association of Supportive Care in Cancer and International Society of Oral Oncology (MASCC/ISOO). MASCC/ISOO clinical practice guidelines for the management of mucositis secondary to cancer therapy. Cancer. 2020 Oct 1;126(19):4423-4431. doi: 10.1002/cncr.33100. Epub 2020 Jul 28. PMID 32786044
- [Result] Cardona A, Balouch A, Abdul MM, Sedghizadeh PP, Enciso R. Efficacy of chlorhexidine for the prevention and treatment of oral mucositis in cancer patients: a systematic review with meta-analyses. J Oral Pathol Med. 2017 Oct;46(9):680-688. doi: 10.1111/jop.12549. Epub 2017 Feb 8. PMID 28075506
- [Result] Ferretti GA, Raybould TP, Brown AT, Macdonald JS, Greenwood M, Maruyama Y, Geil J, Lillich TT, Ash RC. Chlorhexidine prophylaxis for chemotherapy- and radiotherapy-induced stomatitis: a randomized double-blind trial. Oral Surg Oral Med Oral Pathol. 1990 Mar;69(3):331-8. doi: 10.1016/0030-4220(90)90295-4. PMID 2179802